CLINICAL TRIAL: NCT03182257
Title: An Open-label, Multi-center, Dose-escalation and Expansion Study to Evaluate the Safety and Efficacy of ONO-7579 in Patients With Advanced Solid Tumors/ NTRK Gene Fusion Positive Advanced Solid Tumors
Brief Title: Study of ONO-7579 in Patients With Advanced Solid Tumors/ NTRK Gene Fusion Positive Advanced Solid Tumors
Acronym: ONTRK
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped for commercial reasons. No safety issues were reported.
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7579-01
Record Dates: First submitted 2017-05-19; First posted 2017-06-09 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor
Keywords: TRK; TRKA; TRKB; TRKC; NTRK1; NTRK2; NTRK3; NTRK fusion positive; NTRK1 fusion; NTRK2 fusion; NTRK3 fusion; NTRK1 gene rearrangement; NTRK2 gene rearrangement; NTRK3 gene fusion; ETV6-NTRK3; fusion; tumors; solid tumors; CNS tumors; central nervous system tumors; TRK fusion; ETV6; ETV6 fusion; solid CNS tumor; advanced CNS tumor; primary CNS tumor
MeSH Terms: conditions — Neoplasms; Central Nervous System Neoplasms | interventions — ONO-7579

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ONO-7579 Part A (Experimental): Single Ascending doses of ONO-7579
  Interventions: Drug: ONO-7579
- ONO-7579 Part B (Experimental): Expansion phase of ONO-7579
  Interventions: Drug: ONO-7579

INTERVENTIONS:
Drug: ONO-7579 — ONO-7579 Tablets

SUMMARY:
This study will determine the safety and maximum tolerated dose of ONO-7579 in patients with advanced solid tumors, and evaluate efficacy of ONO-7579 in patients with advanced solid tumors harboring NTRK gene fusions.

DETAILED DESCRIPTION:
The trial was designed to be a Phase 1/2 trial, but was terminated without progressing to Phase 2.

ELIGIBILITY:
Inclusion Criteria (Parts A and B):

1. Male or female aged at least 18 years or older, at the time of signing the informed consent form.
2. The patient (or their legal representative) has provided written informed consent, which signifies an agreement to enter the study and comply with the restrictions and requirements listed in the informed consent form.
3. ECOG performance status ≤ 2
4. Life expectancy of at least 3 months
5. Patients must have measurable disease, according to RECIST 1.1 (defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥2 cm) with conventional techniques or as ≥10 mm (≥1 cm) with spiral CT scan), or RANO criteria for Glioma.
6. Patients must have received at least one prior line of therapy appropriate for their tumor type and stage of disease. For glioma, patient must have received at least one prior treatment with radiotherapy and temozolomide. Prior treatment of any Trk inhibitor(s) is not an exclusion.
7. Adequate hematologic, hepatic and renal function as defined by the following criteria:

   * Absolute Neutrophil count ≥ 1.5x109
   * Platelet count ≥ 75,000 / mm3
   * Hemoglobin level ≥ 9.0 g/dL
   * Total Bilirubin level ≤ 1.5 X ULN
   * AST and ALT ≤ 3 X ULN
   * Creatinine clearance* ≥50 mL/min *estimated CLcr by the Cockcroft-Gault equation
8. Women of:

   1. Childbearing potential must have a negative serum pregnancy test documented within 14 days prior to enrollment, and must agree to use two adequate methods of contraception from Day 1 of the study until 3 months after the end of treatment. Acceptable forms of effective contraception include;

      * Established use of oral, injected or implanted hormonal methods of contraception.
      * Placement of an intrauterine device or intrauterine system.
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
      * Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
   2. Non-childbearing potential, defined as females with a documented history of a clinically recognized procedure (e.g. hysterectomy, tubal ligation, bilateral salpingo-/oophorectomy) ; or postmenopausal defined as 12 months of spontaneous amenorrhea with follicle-stimulating hormone (FSH) >40 MlU/mL). Females on hormone replacement therapy (HRT) will be required to use one of the contraception methods in Inclusion criteria 8a or must discontinue HRT to allow confirmation of post-menopausal status prior to being enrolled in the study. Following confirmation of their post-menopausal status, they can resume HRT during the study and will not be required to use contraception.
9. A male patient is eligible to participate if he is not trying to father a child and is willing to use one of the relevant contraception methods as in inclusion criterion 8a from Day 1 of the study until 3 months after the end of treatment.
10. Able to swallow tablets
11. Patients must be recovered to Grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies.

    Additional Criterion for Part A only
12. Patients with histologically/cytologically confirmed advanced solid tumors, and documented tumor progression for whom no further standard anticancer treatment is available.
13. Patients must be able to comply with the protocol requirements regarding fasting, as determined by the investigator (excluding patients in food assessment cohort(s)).

    Additional Criteria for Part B only
14. Patients with histologically/cytologically confirmed advanced solid tumors and documented tumor progression for whom no further standard anticancer treatment exists or where, in the opinion of the investigator, the existing standard anticancer treatment options available are not expected to provide a reasonable benefit to the patient.
15. Patients must have NTRK1, NTRK2 or NTRK3 gene fusion confirmed locally prior to first dose.

Exclusion Criteria:

1. Radiotherapy within two weeks prior to study entry
2. Major surgery (excluding placement of vascular access) within 4 weeks before the first dose of study treatment
3. Spinal cord compression or brain metastases unless treated and radiologically stable for >6 weeks post treatment and not requiring steroids for at least 4 weeks prior to start of study treatment
4. As judged by the Investigator, any evidence of severe or uncontrolled psychiatric disease or systemic diseases, including history of suicide attempt or current suicidal ideation or behavior, active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
5. Concurrent treatment with another investigational agent or participated in another investigational trial within 30 days of study entry
6. Diagnosed or treated for a malignancy other than the tumor under investigation in the study within 5 years, or who were previously diagnosed with a malignancy other than that required for the study and have any radiographic or biochemical marker evidence of that malignancy. Patients with completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy are not excluded.
7. Clinically significant cardiovascular disease, including:

   * History of myocardial infarction, acute coronary syndromes (including unstable angina), or coronary angioplasty/stenting/bypass grafting within the past 6 months.
   * History of Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
   * Severe cardiac arrhythmia requiring medication or other severe conduction abnormalities (e.g. clinically significant QT prolongation or Torsade de pointes)
   * Uncontrolled hypertension
   * Clinically significant valvular disease, cardiomegaly, ventricular hypertrophy, or cardiomyopathy
8. QT prolongation defined as a QTcF interval >470 msec or other significant ECG abnormalities including 2nd degree (type II) or 3rd degree AV block or bradycardia (ventricular rate <50 beats/min) on 12-lead ECG at screening
9. Serious concurrent medical conditions, including serious active infection, in the opinion of the investigator
10. Female patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence, nature and severity of Adverse Events | up to 28 days
  To investigate the safety and tolerability of ONO-7579 to determine MTD/RCD
Part A: Clinically significant changes in physical examinations | up to 28 days
  To investigate the safety and tolerability of ONO-7579 to determine MTD/RCD
Part A: Clinically significant changes in neurological examinations | up to 28 days
  To investigate the safety and tolerability of ONO-7579 to determine MTD/RCD
Part A: Clinically significant changes in vital signs and electrocardiogram - including the evaluation of the QT interval | up to 28 days
  To investigate the safety and tolerability of ONO-7579 to determine MTD/RCD
Part B: Overall Response Rate (ORR) | up to 24 months
  Assessed by Independent Central Review using RECIST 1.1 or RANO criteria

SECONDARY OUTCOMES:
Part A and B Pharmacokinetics (Cmax) | Day 1, 2, 7, 14 and 28
  Assessment of the maximum plasma concentration of ONO-7579
Part A and B Pharmacokinetics (Tmax) | Day 1, 2, 7, 14 and 28
  Assessment of the time to reach maximum observed plasma concentration of ONO-7579
Part A and B Pharmacokinetics (AUC) | Day 1, 2, 7, 14 and 28
  Assessment of the plasma area under the curve from time zero to 24 hours after dosing
Part A and B Pharmacokinetics (T1/2) | Day 1, 2, 7, 14 and 28
  Assessment of the plasma decay half life of ONO-7579
Part A and B Pharmacokinetics (Ctrough) | Day 1, 2, 7, 14 and 28
  Assessment of the trough concentration of ONO-7579 in plasma
Part A Overall Response Rate (ORR) | up to 28 days
  Assessed by investigator using RECIST 1.1 or RANO criteria
Part A Duration of Response (DoR) | up to 28 days
  Assessed by investigator using RECIST 1.1 or RANO criteria
Part A Progression Free Survival (PFS) | up to 28 days
  Assessed by investigator using RECIST 1.1 or RANO criteria
Part B Progression Free Survival (PFS) | up to 24 months
  Assessed by Independent Central Review using RECIST 1.1 or RANO criteria
Part B Overall Survival (OS) | up to 24 months
  Assessed by Independent Central Review using RECIST 1.1 or RANO criteria
Part B Time to Response (TTR) | up to 24 months
  Assessed by Independent Central Review using RECIST 1.1 or RANO criteria
Part B Time to Progression (TTP) | up to 24 months
  Assessed by Independent Central Review using RECIST 1.1 or RANO criteria
Part B Incidence, nature and severity of Adverse Events | up to 24 months
  To determine the safety and tolerability of ONO-7579
Part B: Clinically significant changes in physical examinations | up to 24 months
  To determine the safety and tolerability of ONO-7579
Part B: Clinically significant changes in neurological examinations | up to 24 months
  To determine the safety and tolerability of ONO-7579
Part B: Clinically significant changes in vital signs and electrocardiogram - including the evaluation of the QT interval | up to 24 months
  To determine the safety and tolerability of ONO-7579

CONTACTS AND LOCATIONS:
Overall Officials: Drug Development Division, Study Director — Ono Pharmaceutical Co. Ltd
Locations (5):
- United States (4):
  - Montefiore Medical Center, Lake Success, New York
  - Mount Sinai, New York, New York
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Mary Crowley Cancer Research Center, Dallas, Texas
- Beatson West of Scotland Cancer Centre, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No